CLINICAL TRIAL: NCT03452176
Title: Phase II, Randomized, Single Blind Sham Controlled Trial Investigating Scrambler Therapy for Neuropathic Pain Caused by Neuromyelitis Optica Spectrum Disorder
Brief Title: Scrambler Trial for Pain in NMOSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00115699
Record Dates: First submitted 2018-02-22; First posted 2018-03-02 (Actual); Results first posted 2020-04-17 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Neuromyelitis Optica
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Scrambler (Experimental): This arm will receive the Scrambler intervention for 1 hour daily x10 days.
  Interventions: Device: Scrambler
- Sham-Control (Sham Comparator): This arm will receive the Sham-Control intervention for 1 hour daily x10 days.
  Interventions: Device: Scrambler Sham Control

INTERVENTIONS:
Device: Scrambler — Scrambler is a non-invasive pain modifying technique that utilizes transcutaneous electrical stimulation of nociceptive fibers with the intent of re-organizing maladaptive signaling pathways which has been investigated for treatment of peripheral neuropathy.
  Other Names: CALMARE
  Arms: Scrambler
Device: Scrambler Sham Control — Sham control should be indistinguishable to the participants from experimental Scrambler therapy.
  Arms: Sham-Control

SUMMARY:
A novel technology called Scrambler Therapy is a non-invasive pain modifying technique that utilizes transcutaneous electrical stimulation of C fibers with the intent of re-organizing maladaptive signaling pathways. This neuromodulatory therapy has been investigated for treatment of chronic neuropathic pain in several conditions including chemotherapy-induced peripheral neuropathy, post-herpetic neuralgia and post-surgical neuropathic pain with promising results. Patients report sustained relief after undergoing daily treatment sessions for 10 consecutive weekdays. This study is a randomized single blinded, sham-controlled trial of patients with Neuromyelitis Optica Spectrum Disorder who have central neuropathic pain using Scrambler Therapy added to standardized empiric medications using patient reported outcomes to determine if Scrambler Therapy is a feasible and effective add-on treatment of chronic neuropathic pain.

This trial will recruit twenty-two adult patients diagnosed with NMOSD who have chronic neuropathic pain despite empiric treatment with an anti-epileptic, antidepressant, opioid and/or an NSAID medication. Patients will be randomized 1:1 to undergo Scrambler Therapy or blinded sham daily for 10 days. The primary outcomes will be acceptability and feasibility. The secondary outcome will be efficacy measured as a change in pain scores of more than two points recorded daily by the patient using an 11-point visual analog scale; quality of life (QoL), neurologic function, anxiety, depression, sleep disturbance and pain will also be evaluated at baseline, at the end of therapy, and at 4 & 8 weeks following completion of treatment. Investigators hypothesize that Scrambler Therapy will be an acceptable, feasible and efficacious intervention that significantly reduces pain in patients with neuromyelitis optica spectrum disorder.

DETAILED DESCRIPTION:
Neuromyelitis optica spectrum disorder (NMOSD) is a rare autoimmune disease of the central nervous system that disproportionately affects non-Caucasians and females,1,2 and has a worldwide prevalence estimated to be 0.52 to 4.4/100,000.3 NMOSD preferentially causes recurrent inflammatory attacks in the optic nerves and spinal cord, leading to blindness, paralysis and death. Despite these devastating consequences of the disease, patients have reported that pain is among the most prevalent and debilitating symptom, and impacts mood, mobility and quality of life (QoL). In particular, central neuropathic pain (CNP) is pervasive, severe, intractable to treatment, and affects 62-91% of patients with NMOSD. CNP is described as agonizing burning, stabbing, shooting, tingling or squeezing sensation that is distressing, persistent and incapacitating.13,14 The presence of CNP in NMOSD is a direct consequence of targeted immune-mediated destruction of the spinal cord and may be influenced by lesion span and location: NMOSD lesions are generally transverse, involving both the central gray matter and dorsal horns. The dorsal horns are innervated by primary ascending fibers that convey sensory information to the brain. Damage to the central gray matter in NMOSD leads to astrocytic damage and tissue necrosis, thus disrupting sensory pain tracts going to and from the brain. As a consequence of ongoing spontaneous activity arising in the periphery, surviving neurons develop increased background activity and increased responses to ascending nerve impulses, including normally harmless tactile stimulation. An additional mechanism of CNP involves peripheral sensitization of non-myelinated ascending C fibers interpreted by the brain as persistent pain, a characteristic sign of an inflammatory process in the spinal cord.

Spinal CNP typically presents weeks to months after the cord damage has occurred, long after the acute injury, and may be the result of secondary changes due to reorganization of damaged circuits of the somatosensory system. CNP occurs at and below the spinal cord lesion level, and can persist for years, decades or throughout the patient's life. As with neuropathic pain from other etiologies, the most frequently-used medications for its treatment in NMOSD are anti-epileptics, antidepressants and non-steroidal anti-inflammatory agents. Descriptive studies in NMOSD recognized the inadequate effect of these medications, resulting in frequent breakthrough opioid use. Furthermore, side effects from these medications, particularly at higher doses, are independently associated with fatigue.

Scrambler is a type of transcutaneous electrostimulation (TENS) that uses peripheral nerve stimulation to modify ascending sensory responses in the spinal cord. Electrical impulses are transmitted via surface electrodes placed surrounding the pain area. Traditional TENS units take advantage of the Gate Control Theory in which stimulation of surrounding A-delta fibers dampens incoming pain signals. Scrambler therapy provides additional stimulation of ascending sensory C fibers that imitate normal nerve action potentials with the intent of re-organizing maladaptive signaling pathways. The theory behind Scrambler treatment is that "scrambled" waveforms - instead of repetitive identical waveforms in traditional TENS - are dynamically assembled into strings of information that are interpreted by the brain to replace pain with "no-pain" information. In contrast to traditional TENS therapy that provides only short term pain relief, studies with Scrambler therapy in peripheral neuropathy suggest that patients can have significantly reduced pain or be pain-free for up to 3 months following a series of treatments, and that follow-up treatments may require fewer sessions for continued relief.

This study is a randomized single blinded, sham-controlled trial of patients with Neuromyelitis Optica Spectrum Disorder who have central neuropathic pain using Scrambler Therapy added to standardized empiric medications using patient reported outcomes to determine if Scrambler Therapy is a feasible and effective add-on treatment of chronic neuropathic pain.

This trial will recruit twenty-two adult patients diagnosed with NMOSD who have chronic neuropathic pain despite empiric treatment with an anti-epileptic, antidepressant, opioid and/or an NSAID medication. Patients will be randomized 1:1 to undergo Scrambler Therapy or blinded sham daily for 10 days. The primary outcomes will be acceptability and feasibility. The secondary outcome will be efficacy measured as a change in pain scores of more than two points recorded daily by the patient using an 11-point visual analog scale; quality of life (QoL), neurologic function, anxiety, depression, sleep disturbance and pain will also be evaluated at baseline, at the end of therapy, and at 4 & 8 weeks following completion of treatment. Investigators hypothesize that Scrambler Therapy will be an acceptable, feasible and efficacious intervention that significantly reduces pain in patients with neuromyelitis optica spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Have the presence of persistent CNP rated at a level of 4 or higher on an 11-point numeric rating scale (NRS); persistent pain is defined as presence for >3 months
* Patients must be stable in their disease, such that they have had no spinal cord relapses with the last 6 months
* Patients may use any combination of standard of care medications for pain treatment, to include anti-epileptic, antidepressant, opioid or non-steroidal anti-inflammatory medications, with no adjustments to the regimen within 30 days of enrollment.
* Aquaporin-4 (AQP4)-antibody positive or negative, or untested, but otherwise meeting criteria for diagnosis of NMOSD.

Exclusion Criteria:

* A concomitant diagnosis of peripheral neuropathy
* An ongoing concomitant central neurologic disorder
* Pain that is referable to a spinal cord lesion that starts above the 4th vertebral disc of the cervical spinal cord because FDA device clearance allows for treatment below the neck
* Use of an investigational agent for pain control within 30 days of enrollment
* Pregnant or breastfeeding women
* Those with cognitive or mental incompetency
* Patients with implantable devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levy, MD, PhD, Principal Investigator — Johns Hopkins University; Maureen A Mealy, RN, Study Director — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mealy MA, Kozachik SL, Cook LJ, Totonis L, Salazar RA, Allen JK, Nolan MT, Smith TJ, Levy M. Scrambler therapy improves pain in neuromyelitis optica: A randomized controlled trial. Neurology. 2020 May 5;94(18):e1900-e1907. doi: 10.1212/WNL.0000000000009370. Epub 2020 Apr 8. PMID 32269109

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Scrambler | Sham-Control
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Scrambler | Sham-Control | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean | 56.2 (7.2) | 57.5 (13.8) | 56.9 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Aquaporin-4 Antibody Seropositive [Number; unit: participants] | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Acceptability as Assessed by the Number of Participants Responding Yes to a Question
Description: Will be determined by how many participants say "yes" to the following question, "Would you want to continue the treatment if it were available?"
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Scrambler | Sham-Control
Number analyzed (Participants) | 11 | 11
Participants | 7 | 5

2. Primary Outcome: Feasibility as Assessed by Number of Participants That Completed Treatment Visits
Description: Adherence to visit schedule will be determined by the number of participants that completed the 10 treatment visits.
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Scrambler | Sham-Control
Number analyzed (Participants) | 11 | 11
Participants | 11 | 9

3. Secondary Outcome: Change in Pain Level
Description: Change in NRS pain score (score ranges from 1 to 10 with 1 being "No pain" and 10 being "Worst pain") will be calculated by subtracting the patient's Day 10 pain score (end of treatment) from his or her baseline value.
Time Frame: Baseline, 10 days
Population: Scrambler pre/post compared to sham pre/post using Wilcoxian signed rank
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Scrambler Pre: Median NRS scores prior to receiving 10-day treatment course
- Scrambler Post: Median NRS scores directly following 10-day treatment course to receiving treatment
- Sham Pre: Median NRS scores prior to receiving 10-day sham
- Sham Post: Median NRS scores directly following 10-day sham
Arm/Group | Scrambler Pre | Scrambler Post | Sham Pre | Sham Post
Number analyzed (Participants) | 11 | 11 | 11 | 11
score on a scale | 5.0 [4.25 to 7.0] | 1.5 [0 to 2.75] | 5.0 [4.0 to 7.25] | 4.0 [3.5 to 4.75]

4. Secondary Outcome: Change in Pain Level
Description: as for outcome 3
Time Frame: Baseline, 30 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Scrambler 30-day Post: Median NRS scores 30-day post-treatment
- Sham 30-day Post: Median NRS scores 30-day post sham
Arm/Group | Scrambler 30-day Post | Sham 30-day Post
Number analyzed (Participants) | 11 | 11
score on a scale | 4.5 [3.375 to 5.125] | 5.0 [4.25 to 6.0]

5. Secondary Outcome: Change in Pain Level
Description: as for outcome 3
Time Frame: Baseline, 60 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Scrambler 60-day Post: Median NRS scores 60-day post-treatment
- Sham 60-day Post: Median NRS scores 60-day post sham
Arm/Group | Scrambler 60-day Post | Sham 60-day Post
Number analyzed (Participants) | 11 | 11
score on a scale | 4.5 [2.5 to 5.75] | 5.0 [4.5 to 6.5]

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Scrambler | Sham-Control
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 3/11 | 3/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scrambler (N=11) | Sham-Control (N=11)
Charles Bonnet Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Skin sensitivity to electrodes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 2 (2)
Bacteremia (Infections and infestations) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT03452176/Prot_SAP_000.pdf